CLINICAL TRIAL: NCT06038526
Title: Molecular Studies of Canakinumab in High-Risk Former-Smokers (CANIFS)
Brief Title: Evaluation of Canakinumab in High-Risk Former-Smokers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter Shields (Other)
Responsible Party: Sponsor-Investigator, Peter Shields, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSU-22297; NCI-2023-05942 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-09-06; First posted 2023-09-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cigarette Smoking-Related Carcinoma; Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Specimen Handling; Bronchoscopy; canakinumab; Carbon Monoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (canakinumab, bronchoscopy) (Experimental): Patients undergo bronchoscopy over 30-60 minutes and receive canakinumab SC 60 minutes and 2 weeks after the initial bronchoscopy. Patients undergo an additional bronchoscopy on day 77. Patients undergo buccal, nasal, and blood sample collection and CO testing on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bronchoscopy; Biological: Canakinumab; Procedure: Carbon Monoxide Measurement; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo buccal, nasal, and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bronchoscopy — Undergo bronchoscopy
Biological: Canakinumab — Given SC
  Other Names: ACZ885; Ilaris
Procedure: Carbon Monoxide Measurement — Undergo CO testing
  Other Names: Carbon Monoxide; CO
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase II trial tests the impact of canakinumab on biologic samples (buccal, nasal, and blood) from former smokers with increased risk of cancer. Canakinumab blocks the activity of a protein called interleukin-1 beta (IL-1b), an agent of the inflammatory system and is used for the treatment of different non-cancer diseases (like auto-inflammatory diseases). Giving canakinumab may block the inflammatory system and could have positive effects to reduce cancer growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare baseline bronchoscopy biospecimens with samples approximately 70 days after administration of canakinumab (2 doses, approximately 14 days apart) in healthy former smokers.

SECONDARY OBJECTIVE:

I. Determine the impact of IL-1beta inhibition on downstream inflammatory pathways.

OUTLINE:

Patients undergo bronchoscopy over 30-60 minutes on day 7 and receive canakinumab subcutaneously (SC) 60 minutes and 2 weeks after the initial bronchoscopy. Patients undergo an additional bronchoscopy on day 77. Patients undergo buccal, nasal, and blood sample collection and carbon monoxide (CO testing on study).

ELIGIBILITY:
Inclusion Criteria:

* Age 55-73 (age criteria aligns with Canakinumab Antiinflammatory Thrombosis Outcome Study [CANTOS] trial)
* If female: evidence of post-menopausal status or negative urinary or serum pregnancy test (unknown impact on pregnancy).

Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study treatment and for 6 weeks after stopping medication. Highly effective contraception methods include:

Total abstinence (when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* Male sterilization (at least 6 months prior to screening). For female participants on the study, the vasectomized male partner should be the sole partner for that participant
* Use of oral, (estrogen and progesterone), injected, or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

Women are considered post-menopausal if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age-appropriate history of vasomotor symptoms). Women are considered not of a childbearing potential if they are post-menopausal or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential.

Women will also be considered post-menopausal if they have been amenorrhoeic for 12 months without an alter-native medical cause. The following age-specific requirements apply:

* Women >= 50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)

  * Former smoker with no use in >= 5 years prior to enrollment (targets former smoker population)
  * CO =< 8ppm (targets/confirms former smoker population)
  * Pack-years history of >= 30 (defined as high risk)
  * No unstable or significant medical conditions as determined by medical history (see exclusion criteria below - to ensure safety of the subject, to minimize the effects of poor health on biomarker measures and to maximize compliance to study procedures)
  * C-reactive protein high-sensitivity (hsCRP) levels >= 2 mg/L (defined as increased risk)
  * Negative coronavirus disease (COVID-19) test (if applicable). According to institutional standards, which may evolve throughout the study, if a subject self-reports testing positive for COVID-19, the condition should be resolved without ongoing symptoms for at least three months. If a subject tests positive before the first bronchoscopy, the subject would be placed on a wait list for at least three months and re-tested before his/her appointment; if a subject tests positive before a follow-up bronchoscopy, his/her participation will be withdrawn by the principal investigator (PI)
  * Able to read adequately to complete the survey and related study documents or give consent

Exclusion Criteria:

* Smoked tobacco or cannabis within 5 years of enrollment (target study population is former smokers)
* Used an electronic cigarette or vaped including tetrahydrocannabinol (THC) within 5 years of enrollment (impacts biomarkers). Smoking or vaping any form of tobacco product or cannabis/THC is an exclusion; however, other use of THC administration (e.g., edible, topical, etc.) are permitted
* CO > 8ppm (target study population is former smokers)
* History of or recent exposure to tuberculosis (TB) as documented in the electronic medical record (EMR) and/or testing (impacts risk)
* Body mass index (BMI) > 45 (risk of unstable airway)
* Taking acetylsalicylic acid (ASA) or nonsteroidal anti-inflammatory drugs (NSAIDs) daily or most days per week (impacts biomarkers and risk)
* Concomitant diseases and life-threatening conditions (e.g., cancer or kidney, liver, immune system disorders)
* Prior diagnosis of chronic pulmonary disease (e.g., asthma with regular use of medications, chronic bronchitis, and restrictive lung disease) (impacts biomarkers and risk)
* Acute bronchitis or pneumonia within 1 year (impacts biomarkers)
* COVID-19 diagnosis or related symptoms within the last 3 months (impacts biomarkers and risk). According to institutional standards, which may evolve throughout the study, if a subject self-reports testing positive for COVID-19, the condition should be resolved without ongoing symptoms for at least three months. If a subject tests positive before the first bronchoscopy, the subject would be placed on a wait list for at least three months and re-tested before his/her appointment; if a subject tests positive before a follow-up bronchoscopy, his/her participation will be withdrawn by the PI
* General anesthesia within 1 year (impacts biomarkers)
* Regular use of inhalant medications in the last 3 months (impacts biomarkers)
* Use of antibiotics in prior 30 days (impacts biomarkers)
* Use of steroids, including corticosteroids and inhaled corticosteroids, in prior 30 days (impacts biomarkers)
* Use of prohibited concomitant therapy including but not limited to immunosuppressants (impacts biomarkers and risk). Prohibited concomitant therapy:

  * Immunosuppressants
  * Use of any treatments below is NOT allowed after the start of study treatment due to potential increase in immunosuppressant related concomitant conditions. They are prohibited for the duration of the study and for at least 130 days after discontinuation of study treatment. If a subject chooses to continue one of the medications below, they will be followed.

    * Anti-retro-viral and / or biologic drugs targeting the immune system (e.g., TNF (tumor necrosis factor) blockers, anakinra, rituximab, abatacept, tocilizumab)
    * Immune modulating agent in doses with systemic effects including but not limited to

      * Prednisone > 20 mg (or equivalent) oral or intravenous daily for > 14 days;
      * Prednisone > 5 mg and =< 20 mg (or equivalent) daily for > 30 days;
      * Equivalent dose of methotrexate > 15 mg weekly.
  * Cytochrome P450 Substrates - The formation of CYP450 enzymes is suppressed by increased levels of cytokines (e.g., IL-1) during chronic inflammation. Thus, it is expected that for a molecule that binds to IL-1, such as canakinumab, the formation of CYP450 enzymes could be normalized. This is clinically relevant for CYP450 substrates with a narrow therapeutic index, where the dose is individually adjusted (e.g., warfarin). Upon initiation of canakinumab, in patients being treated with these types of medicinal products, therapeutic monitoring of the effect or drug concentration should be performed and the individual dose of the medicinal product may need to be adjusted as needed
* Live or attenuated vaccines within 90 days of study treatment and after initiation of study drug (impacts biomarkers and risk). Subjects must be discontinued from the trial if administered any live or attenuated vaccine during the course of the study
* Allergies to study medications, such as, lidocaine, versed, fentanyl or cetacaine (impacts risk)
* Bronchoscopy or any other lung procedure for any reason within the previous 6 months (impacts biomarkers)
* Current or recent (within three months) alcohol or drug abuse problems (impacts risk)
* Unable to read for comprehension or completion of study documents (impacts risk)

Ages: 55 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in ASCs (apoptosis-associated speck-like protein containing a caspase activation and recruitment domain) | At baseline and day 77
  Will be assessed by a generalized linear mixed model (GLM) and will be employed with measure as the dependent variable, a main effect of baseline vs. follow-up, covariables sex and age, and a random effect for subject.
Change in caspase-1 | At baseline and day 77
  Will be assessed by a GLM and will be employed with measure as the dependent variable, a main effect of baseline vs. follow-up, covariables sex and age, and a random effect for subject.
Change in interleukin-1 beta (IL-1beta) | At baseline and day 77
  Will be assessed by a GLM and will be employed with measure as the dependent variable, a main effect of baseline vs. follow-up, covariables sex and age, and a random effect for subject.

SECONDARY OUTCOMES:
Changes in immune cell composition in bronchoalveolar lavage (BAL) by mass cytometry (CyTOF) | At baseline and day 77
  Will be performed using SPADE to create a global map of cell types present across samples and how the frequency or activation state of each cell type differs between baseline vs. follow-up (single arm). Will assess batch effects and include batch as a co-variable in the models. Will be assessed by the human magnetic luminex assay on the Luminex platform and inflammatory gene expression by ribonucleic acid sequence (RNASeq).
Changes in cytokines in the blood | At baseline and day 77
  Will be assessed by the human magnetic luminex assay on the Luminex platform and inflammatory gene expression by RNASeq.
Changes in BAL | At baseline and day 77
  Will be assessed by the human magnetic luminex assay on the Luminex platform and inflammatory gene expression by RNASeq.
Bronchoscopy for fractional concentration of exhaled nitric oxide (FeNO) | At baseline and day 77
  Will be assessed by the human magnetic luminex assay on the Luminex platform and inflammatory gene expression by RNASeq.

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Shields, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The James line — http://cancer.osu.edu